CLINICAL TRIAL: NCT06191445
Title: Does the Use of Ultrasound Increase Spinal Anesthesia Success for Obese Patients?: Evaluation of the Success of Spinal Anesthesia Administered with Real-Time Ultrasound-Guided, Ultrasound-Assisted and Conventional Landmark Techniques
Brief Title: Comparison of the Efficacy of Conventional Landmark, Ultrasound-Assisted, and Real-Time Ultrasound-Guided Techniques in Spinal Anesthesia for Obese Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selcan Akesen, Associate Professor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UludagU-KCebeci-002
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Spinal Anesthesia; Ultrasound
Keywords: Anesthesia; Spinal Anesthesia; Obesity; Ultrasonography
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional Landmark Group (Active Comparator): The investigator will perform spinal anesthesia using the conventional landmark technique.
  Interventions: Procedure: Conventional Landmark Technique
- USAS Group (Active Comparator): The investigator will perform spinal anesthesia using ultrasound-assisted technique.
  Interventions: Procedure: Ultrasound Assisted Technique
- US-RTG Group (Active Comparator): The investigator will perform spinal anesthesia using real-time ultrasound-guided technique.
  Interventions: Procedure: Real-Time Ultrasound Guided Technique

INTERVENTIONS:
Procedure: Conventional Landmark Technique — The investigator will perform spinal anesthesia using the conventional landmark technique.
  Arms: Conventional Landmark Group
Procedure: Ultrasound Assisted Technique — The investigator will perform spinal anesthesia using the ultrasound assisted technique.
  Arms: USAS Group
Procedure: Real-Time Ultrasound Guided Technique — The investigator will perform spinal anesthesia using the real-time ultrasound-guided technique.
  Arms: US-RTG Group

SUMMARY:
Spinal anesthesia is frequently administered using the conventional landmark technique. Ultrasound is a non-invasive and safe approach. Neuroaxial anesthesia procedures can be conducted using two different ultrasound techniques; Real-Time Ultrasound Guided (USRTG) and Ultrasound-Assisted (USAS). The primary objective of this study is to compare the successes of spinal anesthesia applications using USRTG, USAS, and conventional landmark techniques on the first attempt in obese patients undergoing orthopedic surgery.

DETAILED DESCRIPTION:
Patients included in the study will be those undergoing lower extremity orthopedic surgery, with a body mass index (BMI) 30 kg/m² and above, and classified as American Society of Anesthesiologists (ASA) class I-III. Patients will be randomized into 3 groups. In the Conventional Landmark group, spinal anesthesia will be administered using the conventional technique. In the Ultrasound-Assisted group, the spinal space will be marked with ultrasound before proceeding. For the Real-Time Ultrasound-Guided group, the spinal space and the advancement of the needle for the injection will be visualized simultaneously with ultrasound during the application of spinal anesthesia. The primary outcome is to compare the success rates on the first attempt. The secondary outcomes are to compare the number of skin punctures, needle redirections, procedure times, complications, and patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patients who will undergo lower extremity orthopedic surgery
* ASA I-II-III patients
* BMI 30 kg/m² and above

Exclusion Criteria:

* BMI < 30 kg/m²
* ASA IV-V patients
* Severe cardiovascular disease
* Patients with a known or suspected allergy to local anesthetics
* Contraindications of spinal anesthesia (eg, coagulopathy, puncture site infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Success rates on the first attempt. | Preoperatively
  The primary outcome is to compare the success rates on the first attempt.

SECONDARY OUTCOMES:
Number of skin punctures, needle redirections, procedure times, complications, and patient satisfaction | Preoperatively
  The secondary outcomes are to compare the number of skin punctures, needle redirections, procedure times, complications (radicular pain, postdural puncture headache, hematoma, paresthesia) and patient satisfaction.
  Needle redirection was defined as any change in needle insertion trajectory not involving complete withdrawal of the needle from the patient's skin.
  Procedure time was defined as the total duration from the placement of the probe on the skin to the completion of skin marking and from the insertion of the needle into the skin to the observation of cerebrospinal fluid (CSF) outflow using the designated technique.
  Patient satisfaction will be evaluated on a scale of 1 to 5 (1:extremely unsatisfied; 5:extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University Faculty of Medicine, Bursa, Turkey (Türkiye)